CLINICAL TRIAL: NCT01223144
Title: Decision-making and Emotion Recognition in Essential Tremor
Acronym: EMOTREM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2010/10
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Essential Tremor
Keywords: Cognition; orbitofrontal cortex; Iowa Gambling Task; facial emotion recognition
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with essential tremor (Experimental): Patients with essential tremor
  Interventions: Behavioral: Iowa Gambling Task and Ekman facial recognition test
- age- and sex-matched control subjects (Active Comparator): age- and sex-matched control subjects
  Interventions: Behavioral: Iowa Gambling Task and Ekman facial recognition test

INTERVENTIONS:
Behavioral: Iowa Gambling Task and Ekman facial recognition test — Iowa Gambling Task: mean number of cards chosen from decks with low (A+B) and high gain (C+D).
  Ekman facial recognition test: mean number of faces correctly recognized (60 images with 6 different expressions: happiness, sadness, fear, surprise, disgust and anger).

SUMMARY:
The present study aims at investigating cognitive functions requiring orbitofrontal control, namely decision-making and facial emotion recognition. The investigators hypothesize that decision-making and facial emotion recognition are impaired in patients with essential tremor (ET) due to frontal lobe dysfunction which may have consequences in daily social life.

DETAILED DESCRIPTION:
Beyond tremor, ET patients display a wide spectrum of clinical abnormalities such as ataxia, deafness, olfactory disturbances, cognitive dysfunction and personality changes. Cognitive dysfunction mainly consists in a dysexecutive syndrome. Personality changes are characterized by increased harm avoidance. These findings suggest a complex modification in frontal lobe function in ET patients, including aspects of dorsolateral and orbitofrontal control. Previous studies have exclusively focused on dorsolateral prefrontal control, while orbitofrontal aspects remain to be elucidated. Orbitofrontal areas are involved in processing emotion and reward, as well as normal social behavior. Dysfunction in these regions may have direct consequences in daily social life.

We hypothesize that decision-making and facial emotion recognition are impaired in ET patients due to frontal lobe dysfunction which may have consequences in daily social life. The first aspect can be assessed with the Iowa Gambling Task, a simple paradigm that simulates real-life decision-making. Briefly, players are given four decks of cards, a loan of $ 2,000 and asked to play so they can lose the least amount of money and win the most. Turning each card carries an immediate reward and sometimes an unpredictable penalty. Decks A and B are the most disadvantageous leading to an overall loss of money, while decks C and D are the most advantageous with an overall gain of money. In contrast to control subjects, patients with damage of the orbitofrontal or ventromedian cortex continue to perseverate with the bad decks, sometimes even though they know that they are losing money overall. The second aspect, i.e. the recognition of facial emotion can be assessed in a simple paradigm where patients have to choose the best fitting response among six facial expressions (happiness, sadness, fear, surprise, disgust and anger) that are presented in random order. All study subjects will be tested with the Benton Visual Retention Test to exclude impairment in visual perception, visual memory or visuoconstructive abilities.

Performances in the Iowa Gambling Task and the facial emotion recognition test will be compared between ET patients and controls. All study subjects will also be tested with the following battery: Modified Card Sorting Test, Stroop, Trail Making Test and Verbal Fluency, Beck Depression Inventory and the Mattis Dementia Rating Scale. These tests will allow assessing the impact of executive function, depression and memory loss on performances in the Iowa Gambling Task and the facial emotion recognition test. Finally, performances in the Iowa Gambling Task and the facial emotion recognition test will be related to sex, age, disease duration and tremor severity.

ELIGIBILITY:
Inclusion Criteria:

* Patient:

  * Age over 18 years
  * Patient diagnosed as having essential tremor
  * Written informed consent
  * Patient covered by the French health insurance system
* Control:

  * Age over 18 years
  * No diagnosis of essential tremor
  * Written informed consent
  * Subject covered by the French health insurance system

Exclusion Criteria:

* Patient:

  * Dementia (MMSE<24) or other known illness which could impact motor and cognitive performances
  * Patient unable to give written informed consent
* Control:

  * Same exclusion criteria as for patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Comparison of the performance in the Iowa Gambling Task and the Ekman facial recognition test | 1 day (duration of study)
  Comparison of the performance in the Iowa Gambling Task and the Ekman facial recognition test between patients and age- and sex-matched controls.
  * Iowa Gambling Task: mean number of cards chosen from decks with low (A+B) and high gain (C+D).
  * Ekman facial recognition test: mean number of faces correctly recognized (60 images with 6 different expressions: happiness, sadness, fear, surprise, disgust and anger).

SECONDARY OUTCOMES:
Risk anticipation as assessed by the number of advantageous minus disadvantageous choices in the Iowa Gambling Task. | 1 day (duration of study)
  Risk anticipation as assessed by the number of advantageous minus disadvantageous choices in the Iowa Gambling Task.
Assessment of the relation between the primary outcome measures and age, sex, disease duration, as well as tremor severity. | 1 day (duration of study)
  Assessment of the relation between the primary outcome measures and age, sex, disease duration, as well as tremor severity.
  Tremor severity is evaluated by the revised WHIGET tremor rating scale (severity score 0-36 points).
Assessment of the relation between the primary outcome measures and executive function and depression. | 1 day (duration of study)
  Executive function Number of categories in the Modified Card Sorting Test Time in seconds and number of errors in the Trail Making Test Time in seconds and number of errors in the Stroop Test Verbal Fluency score Mattis Dementia Rating scale score (0-144 points) Depression is evaluated by the Beck Depression Inventory (0-63 points)

CONTACTS AND LOCATIONS:
Overall Officials: Wassilios Meissner, MD, PhD, Principal Investigator — University Hospital Bordeaux, France
Locations (1):
- CHU de Bordeaux, Hôpital du Haut-Lévêque, Pessac, France